CLINICAL TRIAL: NCT06915467
Title: Efficacy of Direct CAtheterisation of the OMbilical Vein in Emergency Through Wharton's Jelly in the Delivery Room: Multicentre Study
Brief Title: Efficacy of Direct CAtheterisation of the OMbilical Vein in Emergency Through Wharton's Jelly
Acronym: CaDOm
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRD 2419; 2024-515249-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Newborn Morbidity
Keywords: Cardiorespiratory arrest; Newborns; Umbilical Venous Catheter; Wharton's jelly; Neonatal resuscitation; Adrenaline injection
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical vein catheterization through Wharton's jelly (Experimental): All patients included will receive the umbilical route through Wharton's jelly procedure as first-line treatment: placement of the umbilical route through Wharton's jelly, with simultaneous and systematic preparation of umbilical venous catheter (UVC)
  Interventions: Procedure: Umbilical vein catheterization through Wharton's jelly procedure

INTERVENTIONS:
Procedure: Umbilical vein catheterization through Wharton's jelly procedure — All patients included will receive the Umbilical vein catheterization through Wharton's jelly procedure as first-line treatment: placement of the umbilical line through Wharton's jelly, with simultaneous and systematic preparation of umbilical venous catheter (UVC)

SUMMARY:
The aim of this study is to demonstrate, with a good level of evidence, the efficacy, safety and feasibility of placing an umbilical route through Wharton's jelly, in the context of emergency situations in the delivery room.

DETAILED DESCRIPTION:
In France, it is estimated that 2 to 4 births per 1000 are complicated by perinatal anoxia. This infrequent event constitutes a vital emergency because, in addition to death, the consequences, particularly neurological, are serious for the survivors. Mortality is high,and estimated at more than half of children when an Apgar score of zero is observed at 5 and 10 minutes, as shown by data found in the literature. When children are born in circulatory arrest, rapid recovery of a heart rate (HR) of more than 100 beats per minute (bpm) to allow correct circulation is therefore essential.

The recommendations of the European Resuscitation Council, updated in 2021, help to guide the birth room practitioner for optimum effectiveness. If the heart rate remains low, after the ventilation method and interface have been checked and adjusted if necessary, cardiac massage is started, and the next step is the emergency administration of adrenaline via the venous route. The reference route is currently the umbilical venous route via an umbilical venous catheter (UVC). This method is effective, but remains a technical procedure and takes a long time to set up, lasting an average of 3 minutes and up to 6 minutes, including just 1 and a half minutes to prepare the equipment and the venous approach. The intra-tracheal route is not prohibited by the latest recommendations, but it has not been shown to be effective and has not been adopted as a reference emergency route in this indication. The intraosseous route has also been studied and mentioned in the recent recommendations of the Société Française de Néonatalogie, but it remains highly invasive and is not routinely used by neonatal resuscitators or paediatricians in the delivery room. Peripheral venous access is difficult because of hypoperfusion, and is not indicated in these emergency situations either.

In this context, the investigator propose to evaluate a quicker and easier infusion method enabling adrenaline to be administered without delay to neonates in circulatory arrest, when the indication is given, i.e. after a well-conducted initial resuscitation. This method consists of catheterising the umbilical vein directly through Wharton's jelly, and injecting the treatments into it.

The aim of this study is to demonstrate, with a good level of evidence, the efficacy, safety and feasibility of placing an umbilical route through Wharton's jelly, in the context of emergency situations in the delivery room.

ELIGIBILITY:
Inclusion Criteria :

* Full-term newborn (≥ 37 SA)
* Newborn for whom a resuscitation decision has been taken.
* Newborn in circulatory arrest, or in profound bradycardia < 60 bpm, requiring an injection of adrenaline in the delivery room, the indication being established in accordance with the recommendations of the European Resuscitation Council 2021, after completion of the first stages of cardiopulmonary resuscitation, including the establishment of effective ventilation
* Newborn beneficiary of a social security scheme or entitled person.

Non-inclusion Criteria :

* Newborn with known heart defects or other potentially lethal defects
* Presence of a pre-existing access route
* Paediatric resuscitator not trained to the UVW procedure
* Twins born in circulatory arrest and requiring simultaneous management

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Estimation of the success rate of cardiorespiratory resuscitation in less than 90s with the Umbilical vein catheterization through Wharton's jelly as 1st line, in neonates in circulatory arrest in the delivery room | At the beginning of the study, an average of 90 seconds
  Successful completion of the Umbilical vein catheterization through Wharton's jelly procedure is defined as achieving a heart rate (HR) greater than 100 bpm within 90 seconds of the start of the procedure, which corresponds to cord asepsis.
  The reference procedure (UVC), which has been prepared in parallel, is used as soon as it is ready, if the heart rate is not greater than 100 bpm. The Umbilical vein catheterization through Wharton's jelly procedure is then considered to have failed (because the line has not been inserted, the catheter injection has not been performed or the target rate has not been reached within the time limit)

SECONDARY OUTCOMES:
Measurement of the time taken to insert the umbilical line through Wharton's jelly | At the beginning of the study, an average of 90 seconds
  The time taken to insert the umbilical line through Wharton's jelly is the time in seconds between the start of asepsis and the start of catheter injection of adrenaline. To be compared with the time taken to insert the UVC (time between the decision to inject adrenaline and the catheter injection, in order to take into account the time taken to insert the UVC)
Measurement of the delay between the start of the Umbilical vein catheterization through Wharton's jelly procedure and the achievement of a heart rate greater than 100 bpm, to be compared with the delay for an injection via UVC if applicable | At the beginning of the study, an average of 90 seconds
  Delay in seconds between the start of the Umbilical vein catheterization through Wharton's jelly procedure and obtaining a heart rate above 100 bpm, overall and according to the approach actually used (comparison between delay with Umbilical vein catheterization through Wharton's jelly procedure versus UVC procedure where applicable)
Measurement of the delay between the injection of adrenaline by catheter and the resumption of a heart rate greater than 100 bpm, to be compared with the line actually used | At the beginning of the study, an average of 90 seconds
  Delay in seconds between catheter injection of adrenaline and obtaining a heart rate above 100 bpm, overall and according to the approach actually used (comparison between delay with Umbilical vein catheterization through Wharton's jelly procedure versus UVC procedure if applicable)
Measurement of the frequency of failure of the Umbilical vein catheterization through Wharton's jelly procedure | At the beginning of the study, an average of 90 seconds
  The frequency of failure of the Umbilical vein catheterization through Wharton's jelly procedure is the number of failures out of the number of attempts
Description of the types of procedure failure and their causes, requiring the use of another approach | At the beginning of the study, an average of 90 seconds
  The types of failure are: missed deadline, ineffective catheter injection or adverse event.
  Causes of failure may include : a small cord, discoloration/opacity of the cord (icteric or impregnated with meconium), extravasation, failure to locate the vein, absence of reflux, maternal haemorrhage, an equipment-related fault (unsuitable needle, unsuitable syringes), secondary perforation of the vein, inability to keep the needle in the vein during catheter injection, movement of the needle during syringe change for rinsing, or a blood exposure accident (BEA) suffered by the carer
Measurement of immediate mortality (at H1) and mortality at discharge from hospital, or 28 days, overall and according to the approach actually used (Umbilical vein catheterization through Wharton's jelly procedure vs UVC) | At the beginning of the study, an average of 90 seconds
  The mortality rate at H1 and at discharge from hospital (or at 28 days), overall and according to the approach actually used, is the number of patients who died out of the number of patients included
Measurement of tolerance and safety: adverse events within 72 hours, overall and according to the approach used (Umbilical vein catheterization through Wharton's jelly procedure vs UVC) | At 72 hours after the beginning of the study
  Description of adverse events in the 72 hours following catheter injection, overall and according to the approach actually used (Umbilical vein catheterization through Wharton's jelly procedure vs UVC)
Study of the relationship between the delay to inject adrenaline by catheter with the Umbilical vein catheterization through Wharton's jelly procedure and the practitioner's experience, or the condition of the cord | At the beginning of the study, an average of 90 seconds
  Modelling (General Linear Model) of the relationship between, on the one hand, the success or duration of insertion and, on the other hand, the state of the cord (normal or abnormal: if abnormal, it may be thin, meconium-opaque or yellow in the case of jaundice) or the practitioner's experience (number of years ofl experience in neonatal resuscitation and experience of the Umbilical vein catheterization through Wharton's jelly procedure)
Description of the difficulties encountered when using the Umbilical vein catheterization through Wharton's jelly procedure | At the beginning of the study, an average of 90 seconds
  Difficulties encountered during the implementation of this Umbilical vein catheterization through Wharton's jelly procedure will be collected from healthcare professionals and described. These difficulties could be as follows: a lack of confidence on the part of the carer at the time of the procedure, a shortage of staff, difficulty in visualising the vein, an equipment fault (unsuitable needle, unsuitable syringes), an abnormal cord (small, meconium or yellow indicating jaundice), difficulties in keeping the needle in the vein during catheter injection, movement of the needle during the syringe change for rinsing, ...
  Caregivers will also be asked to complete a Likert-type question to assess their feelings about the complexity of the Umbilical vein catheterization through Wharton's jelly procedure. They answer by ticking the box Very easy, Easy, Neither easy nor difficult, Difficult or Very difficult

CONTACTS AND LOCATIONS:
Overall Officials: Dr Suzanne BORRHOMEE, Principal Investigator — Hôpital NOVO - Pontoise site
Locations (5):
- France (5):
  - Paediatric resuscitation and neonatal medicine department- Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Neonatal medicine department - Hôpital Louis Mourier, Colombes
  - Neonatal medicine and resuscitation department - Centre hospitalier intercommunal de Poissy Saint-Germain-en-Laye - Poissy site, Poissy
  - Neonatal medicine - neonatal resuscitation department - Hôpital Delafontaine, Saint-Denis
  - Neonatal medicine and resuscitation department - Centre Hospitalier de Troyes, Troyes